CLINICAL TRIAL: NCT00920855
Title: An Open-Label Study of Bendamustine Combined With Bortezomib for Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Bendamustine Combined With Bortezomib for Patients With Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C18083/1063/MM/US
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Results first posted 2012-09-17 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bendamustine Hydrochloride; Bortezomib

ARMS (1):
- Bendamustine and Bortezomib (Experimental): Bendamustine in escalating doses of 50, 70 or 90 mg/m^2 as combination therapy with bortezomib at 1.0 mg/m^2/dose administered for up to eight 28 day cycles.
  Interventions: Drug: bendamustine; Drug: bortezomib

INTERVENTIONS:
Drug: bendamustine — Bendamustine was administered to 3 cohorts of patients at escalating doses of 50 (cohort 1), 70 (cohort 2) and 90 mg/m^2/dose (cohort 3). Doses were administered by intravenous (iv) infusion once daily on days 1 and 4 of each 28-day cycle. Each iv was administered over 60 minutes and followed the injection of bortezomib.
  Bortezomib will be administered to patients at a dose of 1.0 mg/m2/dose as an iv push over 3 to 5 seconds followed by a standard saline flush or through a running iv line. Doses are to be administered to patients on days 1, 4, 8 and 11 of the 28-day cycle.
  Other Names: CEP-18083; Bendamustine hydrochloride; TREANDA
Drug: bortezomib — Bortezomib was administered at a dose of 1.0 mg/m^2/dose as an intravenous (iv) push over 3 to 5 seconds followed by a standard saline flush or through a running iv line. Doses are to be administered on days 1, 4, 8 and 11 of each 28-day cycle.
  Other Names: VELCADE®

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of bendamustine as combination therapy with bortezomib for patients with relapsed/refractory multiple myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

The patient:

* has a diagnosis of multiple myeloma.
* currently has multiple myeloma with measurable disease.
* must have received at least 1 previous treatment regimen and shows signs of progressive disease at the time of study entry.
* if a woman of child bearing potential (not surgically sterile or at least 12 months naturally postmenopausal), must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study.
* if a man, must agree to use an acceptable method of contraception throughout the study and for 90 days after last dose study drug.
* must have an Eastern Cooperative Oncology Group (ECOG) performance status not greater than 2.
* must have a life-expectancy of greater than 3 months.
* must meet specific protocol-related hematological and laboratory criteria within 14 days of enrollment.

Exclusion Criteria:

The patient has:

* had a prior malignancy within the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix).
* plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes (POEMS) syndrome.
* plasma cell leukemia.
* non-measurable multiple myeloma.
* Common Terminology Criteria for Adverse Events (CTCAE) grade 2 (or greater) peripheral neuropathy within 14 days before enrollment.
* previously participated in a Cephalon-sponsored clinical study with bendamustine.
* impaired cardiac function or clinically significant cardiac diseases.
* undergone major surgery within 4 weeks prior to screening or has not recovered from side effects of such therapy.
* severe hypercalcemia.
* other concurrent severe and/or uncontrolled medical or psychiatric conditions.
* known positivity for human immunodeficiency virus (HIV) or hepatitis B or C.
* a history of allergic reaction attributable to compounds of similar chemical or biological composition to bendamustine, bortezomib, boron, or mannitol.
* received chemotherapy within 3 weeks before enrollment, with the exception of nitrosoureas, which should be discontinued at least 6 weeks before enrollment.
* received corticosteroids (greater than 10 mg/day prednisone or equivalent) within 3 weeks before enrollment.
* received immunotherapy, antibody, or radiation therapy within 4 weeks before enrollment.
* a status as a pregnant or lactating woman. Any women becoming pregnant during the study will be withdrawn from the study.
* a status as a male whose sexual partner is a woman of childbearing potential not using effective birth control.
* used an investigational drug within 1 month before the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon
Locations (13):
- United States (13):
  - Pacific Oncololgy & Hematology, Encinitas, California
  - Capitol Hematology Oncology, Roseville, California
  - University Of California, San Diego, San Diego, California
  - James R. Berenson, M.D., Inc., West Hollywood, California
  - George Washington University, Washington D.C., District of Columbia
  - Northshore University Health System, Evanston, Illinois
  - Alivin & Lois Lapidus Cancer Institute, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Sophia Gordon Cancer Center at Lahey Clinic, Burlington, Massachusetts
  - Geisinger Medical Center, Danville, Pennsylvania
  - Charleston Hematology Oncology, PA, Charleston, South Carolina
  - Family Cancer Center, PLLC, Collierville, Tennessee
  - Fairfax Northern Virginia Hematology Oncology, Fairfax, Virginia

REFERENCES:
- [Result] Berenson JR, Yellin O, Bessudo A, et al. Bendamustine combined with bortezomib has efficacy in patients with relapsed or refractory multiple myeloma: a phase 1/2 study. Blood (ASH Annual Meeting Abstracts). 2011;118 (suppl 21):abstract 1857

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifty-one patients were screened and forty from 10 U.S. centers were enrolled. Reasons for not enrolling were failed to meet inclusion and/or exclusion criteria (10) and an adverse event (1).
Groups:
- Bendamustine 50 mg/m^2 Cohort: Bortezomib 1.0 mg/m^2/dose (days 1, 4, 8 and 11) by intravenous push and Bendamustine 50 mg/m^2/dose (days 1 and 4) intravenously for up to eight 28 day cycles.
- Bendamustine 70 mg/m^2 Cohort: Bortezomib 1.0 mg/m^2/dose (days 1, 4, 8 and 11) by intravenous push and Bendamustine 70 mg/m^2/dose (days 1 and 4) intravenously for up to eight 28 day cycles.
- Bendamustine 90 mg/m^2 Cohort: Bortezomib 1.0 mg/m^2/dose (days 1, 4, 8 and 11) by intravenous push and Bendamustine 90 mg/m^2/dose (days 1 and 4) intravenously for up to eight 28 day cycles.
Period: Overall Study
Arm/Group | Bendamustine 50 mg/m^2 Cohort | Bendamustine 70 mg/m^2 Cohort | Bendamustine 90 mg/m^2 Cohort
Started | 5 | 4 | 31
Safety and Efficacy Populations | 5 | 4 | 31
Completed | 0 (completed eight cycles of treatment) | 1 (completed eight cycles of treatment) | 9 (completed eight cycles of treatment)
Not Completed | 5 | 3 | 22
Not completed — Adverse Event | 1 | 1 | 4
Not completed — Withdrawal by Subject | 2 | 1 | 6
Not completed — Disease progression | 2 | 1 | 10
Not completed — Noncompliance to study medication | 0 | 0 | 1
Not completed — Response plateau; started maintenance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bendamustine 50 mg/m^2 Cohort | Bendamustine 70 mg/m^2 Cohort | Bendamustine 90 mg/m^2 Cohort | Total
Number analyzed (Participants) | 5 | 4 | 31 | 40
Age Continuous [Mean (Standard Deviation); unit: years] | 62.8 (18.17) | 67.0 (9.49) | 64.5 (10.68) | 64.6 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 12 | 17
  Male | 2 | 2 | 19 | 23
Race/Ethnicity, Customized [Number; unit: participants]
  White | 4 | 4 | 24 | 32
  Black | 1 | 0 | 5 | 6
  Asian | 0 | 0 | 1 | 1
  Other | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 31 | 40
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.76 (0.234) | 1.81 (0.177) | 1.90 (0.265) | 1.87 (0.254)

OUTCOME MEASURES:

1. Primary Outcome: Participants With Dose Limiting Toxicity (DLT)
Description: Maximum tolerated dose was the dose that was 1 step lower than the dose where at least one third of patients experienced DLT. A DLT was defined as any of the following occurring during the first cycle:
  * grade 4 hematologic toxicity without regard for relationship to study drug treatment
  * thrombocytopenia grade 3 with grade 3 or grade 4 hemorrhage
  * grade 3 febrile neutropenia
  * grade 3 or grade 4 nausea and vomiting refractory to anti emetic therapy
  * any study drug related grade 3 or grade 4 nonhematologic toxicity
  * any drug related death
  Toxicity grades (3=severe AE and 4=life-threatening or disabling AE) were assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.
Time Frame: Day 1 - 28
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Bendamustine 50 mg/m^2 Cohort | Bendamustine 70 mg/m^2 Cohort | Bendamustine 90 mg/m^2 Cohort
Number analyzed (Participants) | 5 | 4 | 31
participants | 0 | 0 | 0

2. Secondary Outcome: Percentage of Participants With An Overall Tumor Response As Assessed By the Investigator
Description: Overall tumor response is the sum of a complete response (CR), very good partial response (VGPR), partial response (PR) and minimal response (MR). A modified version of the Bladé criteria for response was used. Abbreviated definitions for the response categories can be found in the description of outcome #3.
Time Frame: Up to 7.5 months (eight 28-day cycles)
Population: Efficacy population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine 50 mg/m^2 Cohort | Bendamustine 70 mg/m^2 Cohort | Bendamustine 90 mg/m^2 Cohort
Number analyzed (Participants) | 5 | 4 | 31
percentage of participants | 40.0 [5.27 to 85.34] | 25.0 [0.63 to 80.59] | 51.6 [33.06 to 69.85]

3. Secondary Outcome: Participants' Best Tumor Response as Assessed by the Investigator
Description: Abbreviated criteria for response categories: CR includes the disappearance of the original monoclonal protein (M-protein) from blood and urine, and <5% plasma cells in the bone marrow, and no increase in size/number of lytic bone lesions, and disappearance of soft tissue plasmacytomas for >=4 weeks. VGPR includes serum and urine M-protein detectable by immunofixation but not electrophoresis, and reduction in 24-hr urinary light chain excretion by <100 mg, and disappearance of soft tissue plasmacytomas for >= 4 weeks, and no increase in size/number of lytic bone lesions. PR includes a >=50% reduction in serum M-protein, and reduction in 24-hr urinary light chain excretion by either >=90% or to <200 mg, and >=50% reduction in size of soft tissue plasmacytomas, and no increase in size/number of lytic bone lesions. MR includes a >=25% and <=49% reduction in serum M-protein. SD does not meet criteria for the other response categories. See outcome #4 for a definition of PD.
Time Frame: up to 7.5 months (eight 28-day cycles)
Population: Efficacy population
Measure: Number; unit: participants
Arm/Group | Bendamustine 50 mg/m^2 Cohort | Bendamustine 70 mg/m^2 Cohort | Bendamustine 90 mg/m^2 Cohort
Number analyzed (Participants) | 5 | 4 | 31
participants
  Complete response (CR) | 0 | 0 | 1
  Very good partial response (VGPR) | 0 | 0 | 2
  Partial response (PR) | 1 | 0 | 8
  Minimal response (MR) | 1 | 1 | 5
  Stable disease (SD) | 2 | 2 | 13
  Progressive disease (PD) | 1 | 1 | 2

4. Secondary Outcome: Kaplan-Meier Estimate for Time to Progression (TTP)
Description: Time to progression was defined as the time from initiation of therapy to progressive disease (PD). PD requires at least one of the following:
  * >25% increase in serum monoclonal paraprotein (which must also be an absolute increase of at least 5 g/L),
  * >25% increase in 24-hour urinary light chain excretion (which must also be an absolute increase of at least 200 mg/24 h),
  * >25% increase in plasma cells in a bone marrow aspirate or on trephine biopsy (which must also be an absolute increase of at least 10%),
  * definite increase in the size of existing lytic bone lesions or soft tissue plasmacytomas,
  * the development of new bone lesions or soft tissue plasmacytomas,
  * the development of hypercalcemia (corrected serum calcium > 11.5 mg/dL or 2.8 mmol/L not attributable to any other cause).
Time Frame: up to 8.6 months
Population: Safety population
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bendamustine and Bortezomib - Overall: Bendamustine in escalating doses of 50, 70 or 90 mg/m^2 as combination therapy with bortezomib at 1.0 mg/m^2/dose administered for up to eight 28 day cycles. Participants whose disease has not progressed at the end of the eight cycles will be followed until disease progression or death.
Arm/Group | Bendamustine and Bortezomib - Overall
Number analyzed (Participants) | 40
months | 8.4 [4.03 to NA] — Upper boundary was not estimated due to the limited number of participants with events.

5. Secondary Outcome: Kaplan-Meier Estimate for Progression-Free Survival
Description: Progression free survival is the time between the date of initiation of therapy to progressive disease (PD) or death from any cause, whichever occurs first. See outcome #4 for a definition of PD.
Time Frame: up to 23 months
Population: Safety population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine and Bortezomib - Overall
Number analyzed (Participants) | 40
months | 15.21 [5.22 to 16.63]

6. Secondary Outcome: Time to the First Response
Description: Time to first response is defined as the time from the initiation of therapy to the first evidence of a confirmed response (ie, CR, VGPR, PR, or MR).
Time Frame: up to 8.5 months
Population: Participants who had a response
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Bendamustine and Bortezomib - Overall
Number analyzed (Participants) | 19
months | 1.9 (1.51)

7. Secondary Outcome: Kaplan-Meier Estimate for Duration of Response
Description: Duration of response (DR) is defined as the time from the first response to progressive disease (PD). See outcome #4 for a PD definition.
Time Frame: up to 8.5 months
Population: Participants who had a response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine and Bortezomib - Overall
Number analyzed (Participants) | 19
months | NA [6.55 to NA] — Median and upper boundary were not estimated due to the limited number of participants with events.

8. Secondary Outcome: Kaplan-Meier Estimate for Overall Survival (OS)
Description: Overall survival is defined as the time from initiation of therapy to death from any cause or last follow-up visit.
Time Frame: up to 23 months
Population: Safety population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine and Bortezomib - Overall
Number analyzed (Participants) | 40
months | 17.82 [15.83 to NA] — Upper boundary was not estimated due to the limited number of participants with events.

9. Secondary Outcome: Summary of Participants With Adverse Events (AEs)
Description: Counts of participants who had AEs are summarized in a variety of categories. Severity and relatedness to study drug are in the opinion of the investigator according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0. Severity is rated on a 5-point scale: 1=mild, 2=moderate, 3=severe, 4=life threatening or disabling, and 5= death related to AE. Relatedness is assessed on a 5-point scale: not related, unlikely, possible, probable and definite. Definite, probable and possible answers are reported as 'related' to study medication. Deaths are reported up to 18 months. All the deaths occurred beyond the treatment-emergent timeframe since they occurred 6.5-16 months after the final dosing. All other parts of the summary represent the treatment-emergent timeframe (up to 8.5 months) which is the treatment period plus 30 days.
Time Frame: up to 8.5 months. Deaths are reported up to 18 months
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Bendamustine 50 mg/m^2 Cohort | Bendamustine 70 mg/m^2 Cohort | Bendamustine 90 mg/m^2 Cohort
Number analyzed (Participants) | 5 | 4 | 31
participants
  Any adverse event | 5 | 4 | 31
  Any non-haematologic adverse event | 5 | 4 | 31
  Severe adverse event (grade 3 or 4) | 3 | 3 | 22
  Treatment-related adverse events | 4 | 4 | 31
  Deaths | 1 | 0 | 5
  Serious adverse events | 0 | 1 | 7
  Withdrawn from study due to AE | 2 | 2 | 5

ADVERSE EVENTS:
Time Frame: up to 8.5 months
Arm/Group | Bendamustine 50 mg/m^2 Cohort | Bendamustine 70 mg/m^2 Cohort | Bendamustine 90 mg/m^2 Cohort
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/4 | 7/31
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bendamustine 50 mg/m^2 Cohort (N=5) | Bendamustine 70 mg/m^2 Cohort (N=4) | Bendamustine 90 mg/m^2 Cohort (N=31)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 2
Cystitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Sepsis syndrome (Infections and infestations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bendamustine 50 mg/m^2 Cohort (N=5) | Bendamustine 70 mg/m^2 Cohort (N=4) | Bendamustine 90 mg/m^2 Cohort (N=31)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 19
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 10
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 15
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0
Scleral hyperaemia (Eye disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 11
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 9
Nausea (Gastrointestinal disorders) | 1 | 3 | 21
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 10
Fatigue (General disorders) | 3 | 4 | 17
Infusion site irritation (General disorders) | 1 | 0 | 0
Local swelling (General disorders) | 1 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 2
Chills (General disorders) | 0 | 0 | 2
Influenza like illness (General disorders) | 0 | 0 | 3
Oedema peripheral (General disorders) | 0 | 1 | 5
Pain (General disorders) | 0 | 1 | 2
Pyrexia (General disorders) | 0 | 0 | 6
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Nail bed infection (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 9
Catheter site cellulitis (Infections and infestations) | 0 | 1 | 0
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 0 | 6
Pneumonia (Infections and infestations) | 0 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 4
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Haemoglobin decreased (Investigations) | 1 | 3 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Blood calcium decreased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 4
Blood glucose increased (Investigations) | 0 | 0 | 2
Blood magnesium decreased (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 2
Hematocrit decreased (Investigations) | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 0 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 11
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Muscularskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Muscularskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 5
Neuropathy peripheral (Nervous system disorders) | 1 | 2 | 10
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 4
Paraesthesia (Nervous system disorders) | 0 | 0 | 3
Tremor (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 4
Breast tenderness (Reproductive system and breast disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 2
Vein pain (Vascular disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.